CLINICAL TRIAL: NCT01389687
Title: Immunogenicity and Safety of the SP059 Given Subcutaneously as a Three-dose Primary and Booster Vaccination in Infants in Japan
Brief Title: Study of SP059 Given Subcutaneously as a Three-dose Primary and Booster Vaccination in Infants in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPV35 (EFC12403); U1111-1120-1735 (Other: WHO)
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Poliomyelitis; Polio
Keywords: Poliomyelitis; Inactivated polio vaccine; Polio; Poliovirus
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Biological: Inactive Poliovirus Vaccine

INTERVENTIONS:
Biological: Inactive Poliovirus Vaccine — 0.5 mL, Subcutaneous
  Other Names: SP059

SUMMARY:
The aim of the study is to assess the immunogenicity and safety of SP059 as a three-dose primary and booster vaccination in Japanese infants aged 3 through 68 months.

Primary objective:

* To assess that the seroprotection rates against polio types 1, 2 and 3 are over 90% approximately one month following the three dose primary vaccination series with inactivated polio vaccine (IPV).

Secondary objective:

* To describe the immunogenicity (in terms of seroprotection / seroconversion vaccine response rates and Geometric Mean Titers) of IPV before and after the primary vaccination and before and after the booster vaccination.
* To describe the safety after each dose of IPV.

DETAILED DESCRIPTION:
Study participants will receive three doses of inactivated polio vaccine (IPV) (at each visit and given 3-8 weeks apart) as a three-dose primary vaccination starting at 3-68 months of age and followed by a single dose of IPV as a booster vaccination 6-18 months after completion of the three-dose primary vaccination.

Subjects will be observed by the Investigator or sub-Investigator for 30 minutes following the vaccine injection.

The duration of each participant's participation in the trial will be approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 to 68 months inclusive (recommended 3 to 8 months) on the day of inclusion
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures Exclusion Criteria:
* Fever ≥ 37.5°C (axillary temperature) on the day of inclusion
* Any serious disease whether acute or chronic
* History of poliomyelitis infection
* History of a life threatening reaction to a vaccine containing the same substances of the study vaccine
* History of anaphylaxis or allergy to any of the study vaccine components
* Previous vaccination against the poliomyelitis diseases infection with a trial vaccine or another vaccine
* Congenital or current/ previous acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy
* Participation in another clinical trial preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Blood or blood-derived products received in the past or current or planned administration during the trial (including immunoglobulins).
* Any vaccination with live vaccines within the past 27 days preceding the first trial vaccination.
* Any vaccination with inactivated vaccines within the past 6 days preceding the first trial vaccination.
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or human immunodeficiency virus infection
* Subject ineligible according to the investigator's clinical judgment.

Ages: 3 Months to 68 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
A description of the anti-Polio 1, 2 and 3 antibody titers post-vaccination | 1 month post-vaccination 3
  Anti-Polio 1, 2 and 3 antibody titers will be determined by the Seroneutralization assay.

SECONDARY OUTCOMES:
Immunogenicity (in terms of seroprotection and Geometric Mean Titers) of inactivated polio vaccine (IPV) before and after the primary vaccination and before and after the booster vaccination. | Day 0 and 1 month post-vaccination
Description of the safety profile in terms of solicited injection site and systemic reaction, and serious adverse events after each vaccination with IPV | Day 0 up to 12 months post-vaccination
  Solicited injection site: Tenderness (3 to 23 months); Pain (2 to 11 years), Redness, and Swelling. Solicited Systemic reaction: 3 to 23 month olds: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of Appetite, and Irritability: 2 to 11 year olds: Fever (Temperature), Headache, Malaise, and Myalgia.
Immunogenicity (in terms of anti-Polio 1, 2, and 3 titers ≥ 8 [1/dilution], individual antibodies' titers and Geometric Mean Titers) of inactivated polio vaccine (IPV) after the booster vaccination. | 1 month post-booster vaccination
  Anti-Polio 1, 2 and 3 antibody titers will be determined by the Seroneutralization assay.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Aventis K.K.
Locations (2):
- Japan (2):
  - Fukui-shi, Fukui
  - Sapporo, Hokkaido

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com